CLINICAL TRIAL: NCT00236470
Title: Risperidone in the Treatment of Children and Adolescents With Conduct and Other Disruptive Behavior Disorders - an Open Label Follow-up Trial of CR002020
Brief Title: A Study of the Safety of Risperidone in the Treatment of Children and Adolescents With Conduct and Other Disruptive Behavior Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002149
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Disruptive Behavior Disorder
Keywords: Disruptive behavior disorder; risperidone; antipsychotropic agents; child; adolescent
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The primary purpose of this study is to document the long-term safety of an oral formulation of risperidone in the treatment of children and adolescents with conduct and other disruptive behavior disorders. Data on the efficacy of the drug will also be collected. Only patients who were enrolled in the previous related study would be eligible to participate.

DETAILED DESCRIPTION:
This is an open-label study of an oral formulation of risperidone to be taken daily over 12 months by children and adolescents with conduct and other disruptive behavior disorders. It is an extension of a randomized, double-blind study (RIS-INT-79) comparing risperidone with placebo over 6 months in patients who had already shown response to the medication for a period of 12 weeks. Efficacy assessments include: the Conduct Problem subscale of the Nisonger Child Behavior Rating Form (N-CBRF), a measure of symptoms of conduct and other disruptive behavior disorders; Visual Analogue Scale for the most troublesome symptom (VAS-MS), a scale ranging from not troublesome to extremely troublesome; Clinical Global Impression-Severity of Illness (CGI-Severity), a measure of overall severity of illness; Children's Global Assessment Scale (C-GAS), as assessment overall functioning. Safety evaluations include incidence of adverse events, physical examinations, laboratory tests (biochemistry, hematology, and urinalysis), and electrocardiograms (ECGs). Oral risperidone solution (1milligram/milliliter) daily for 1year. For patients weighing at least 50kg, start dose is 0.5ml/day. At investigator's discretion, dose may be increased (maximum 1.5ml/d over 5 days). Patients under 50kg start at 0.25ml/d, increased, if required, to maximum 0.75ml/d.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the double-blind study (CR002020)
* Patients must begin the present study within 7 days of taking the last dose of medication in the prior study (CR002020)

Exclusion Criteria:

* Patients with hypersensitivity or intolerance to risperidone
* Patients with extrapyramidal symptoms (EPS) not adequately controlled with medication
* History of neuroleptic malignant syndrome, a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness
* Significant and untreated or unstable medical illness such as diabetes, hypertension
* serious illness of the liver, kidney, or significant disturbances of the cardiac, pulmonary, gastrointestinal, endocrine, neurological system
* Pregnant or nursing females, or those lacking adequate contraception

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 232 (Actual)
Dates: Start 2002-01; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
To accumulate long-term safety data: incidence of adverse events and clinical evaluations (physical exam, laboratory tests) conducted throughout the trial.

SECONDARY OUTCOMES:
To asses long-term efficacy data: changes from baseline to 1 year in Conduct Problem subscale of N-CBRF; VAS-MS changes from baseline through 1 year; CGI-Severity subscale at every visit; C-GAS rated for global functioning at the endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the safety of risperidone in the treatment of children and adolescents with conduct and other disruptive behavior disorders — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=452&filename=CR002149_CSR.pdf